CLINICAL TRIAL: NCT04919096
Title: A Phase 1, Randomized, Double-Masked, Parallel Group, Multicenter, Pilot Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SCB-420 and Eylea® in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: Study of SCB-420 in Subjects With Neovascular Age-related Macular Degeneration
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to an internal decision to prioritise its development pipeline, Clover have decided to close down study CLO-SCB-420-001. This was a corporate decision and not the results of new data or information arising related to SCB-420
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLO-SCB-420-001
Record Dates: First submitted 2021-05-18; First posted 2021-06-09 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Wet Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCB-420 (Experimental): Subjects randomized to SCB-420 will receive SCB-420 2mg (0.05 mL) via intravitreal injection in the study eye every 4 weeks for the first 3 months.
  Interventions: Drug: SCB-420
- Aflibercept (Active Comparator): Subjects randomized into Aflibercept (Eylea) group will receive Aflibercept (Eylea) 2 mg (0.05 mL) via intravitreal injection in the study eye every 4 weeks for the first 3 months.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: SCB-420 — Subjects randomised to SCB-420 arm will receive a total of 3 doses of SCB-420 as an intravitreal injection of 2 mg into the study eye every 4 weeks on Day 1, Week 4, and Week 8.
  Arms: SCB-420
Drug: Aflibercept — Subjects randomised to Aflibercept arm will receive a total of 3 doses of Aflibercept as an intravitreal injection of 2 mg into the study eye every 4 weeks on Day 1, Week 4, and Week 8.
  Other Names: Eylea
  Arms: Aflibercept

SUMMARY:
This is a Phase 1, randomized, double-masked, multicenter, parallel-assignment, pilot study to evaluate the safety, tolerability, initial clinical effectiveness, pharmacokinetics (PK), and immunogenicity of SCB-420 as compared with Eylea (aflibercept), in subjects with Neovascular Age-related Macular Degeneration.

A total of 20 subjects with Neovascular Age-related Macular Degeneration will be enrolled across up to 11 sites in 3 countries (Australia, New Zealand, and China). The study will be conducted in 2 parts - Sentinel Safety Cohort and Open Enrolment. Subjects will be administered with 2 mg of SCB-420 or Eylea via intravitreal (IVT) injection every 4 weeks for a total 3 doses.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 50 years of age.
2. Willing and able to provide written informed consent prior to any study procedure. Willing and able to comply with all protocol requirements, schedules, and procedures.
3. Treatment-naïve, active choroidal subfoveal neovascularization lesions secondary to Age-related Macular Degeneration (AMD) evidenced by Fluorescein Angiography (FA) and Indocyanine Green Angiography (ICGA) (including PCV) in the study eye evidenced by subfoveal FA/ICGA leakage, or definite subfoveal fluid by spectrum domain optical coherence tomography (SD-OCT) at screening by the Study Doctor but confirmed by the independent image reading center.

   1. Active Choroidal neovascularization (CNV) area occupies at least 50% of the total lesion area in the study eye.
   2. Total lesion area (including blood, scars, and vascularization) is ≤9.0 Disc Areas (DA) in the study eye.
4. Best corrected visual acuity (BCVA) letter score of 78 to 25 inclusive, using Early Treatment Diabetic Retinopathy Study (ETDRS) charts or 2702 series number charts in the study eye at screening and at Day 1 prior to randomization (20/32 to 20/320 Snellen equivalent). The fellow (non-study) eye should not have BCVA letter score less than 19 letters (20/400 Snellen equivalent).
5. Women of childbearing potential with a negative serum pregnancy test at screening must agree to use protocol-defined methods of contraception for 30 days prior to the first dose of the study and throughout the study until 3 months after the last injection of Eylea or SCB-420.
6. Males with female partners of childbearing potential must agree to use protocol-defined methods of contraception and agree to refrain from donating sperm throughout the study until 3 months after the last injection of Eylea or SCB-420.
7. Have ocular media (lens, cornea, vitreous) of adequate clarity to permit high quality fundus imaging.

Exclusion Criteria:

Study Eye

1. Sub- or intra-retinal hemorrhage that comprises more than 50% of the entire lesion or presence of blood with the size of 1 Disc Areas (DA) or more involving the center of fovea.
2. Have scarring or fibrosis making up greater than 50% of total lesion in the study eye at screening; and/or scarring, fibrosis or atrophy involving the center of the fovea in the study eye at screening.
3. Choroidal neovascularization due to other causes, such as ocular histoplasmosis, trauma, punctate inner choroidopathy/multifocal choroiditis, angioid streaks, history of choroidal rupture, or pathologic myopia.
4. History of macular hole of Stage 2 and above.
5. Macular pathology other than Age-related Macular Degeneration that might compromise central vision, i.e., vitreomacular traction or significant epiretinal membrane. Polypoid choroidal vasculopathy identified on screening ICGA is not exclusionary.
6. Presence of retinal pigment epithelial tears or rips involving the macula.
7. History of any vitreous hemorrhage in the study eye within 8 weeks prior to the screening visit.
8. History of retinal detachment, treatment, or surgery for retinal detachment in the study eye.
9. Uncontrolled ocular hypertension (defined as Intraocular Pressure (IOP) ≥22 mmHg despite treatment with anti-glaucoma medication) at screening.
10. Significant media opacities, including Lens Opacities Classification System (LOCS) II Grade IV cataract in the study eye, or other significant cataract in the study eye that in the investigator's opinion interferes with visualization of retina or interferes with retinal imaging.
11. Aphakia or absence of the posterior capsule (unless it occurred as a result of a yttrium aluminum garnet (YAG) laser posterior capsulotomy in association with prior posterior chamber Intraocular Lens (IOL) implantation) in the study eye.
12. History or evidence of any other clinically significant disorder, condition or disease (e.g., co-existence of retinal vein occlusion (RVO), radiation retinopathy, diabetic retinopathy, glaucoma under treatment) in the study eye that, in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedure or complication.
13. Have active intraocular inflammation in either eye at screening or upon examination at baseline or a history of uveitis in either eye.
14. Have active ocular or periocular infection in either eye, or a history of any ocular or periocular infection within the 2 weeks prior to screening in either eye.

    Study Eye - Ocular Treatment/Surgical History
15. Any prior ocular or systemic treatment, surgery, or investigational product for neovascular Age-related Macular Degeneration, including anti-vascular endothelial growth factor (anti-VEGF) therapy, except dietary supplements or vitamins.
16. Prior treatment with intravitreal (IVT) anti-VEGF therapy for any other indication.
17. Have participated as a subject in any interventional clinical trial within 1 month (30 days) prior to the baseline visit.
18. History of vitrectomy or treatment of the macula with verteporfin (photodynamic therapy), transpupillary thermotherapy, radiation therapy, or retinal laser treatment (e.g., focal laser photocoagulation) in the study eye.
19. History of laser therapy of the macula.
20. History of glaucoma-filtering surgery within 3 months of Day 1 in the study eye. Anti-glaucoma laser surgeries are allowed.
21. History of corneal transplant or presence of a corneal dystrophy that interferes with intraocular pressure measurements or imaging in the study eye.
22. Any other intraocular or periocular surgery within 3 months prior to Day 1. Lid surgery prior to 1 month of Day 1 is allowed. Uncomplicated neodymium-doped yttrium aluminium garnet (Nd:YAG) laser capsulotomy performed for secondary opacification of the posterior capsule in IOL-implanted eye within 3 months prior to Day 1 is allowed.
23. History of intravitreal or periocular injections of corticosteroids within 6 months prior to screening in the study eye or device implantation in the prior 36 months.
24. Have any use of long acting intraocular steroids, including implants, within 6 months prior to Day 1, baseline.

    Either Eye
25. History or clinical evidence of diabetic retinopathy, diabetic macular edema (DME), or any other vascular disease affecting the retina, other than Age-related Macular Degeneration in either eye.
26. Active intraocular inflammation or active or suspected ocular or periocular infection, within 2 weeks before Day 1.
27. Active scleritis or episcleritis or presence of scleromalacia.

    Other
28. Uncontrolled hypertension defined as systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg under appropriate antihypertensive treatment.
29. Thrombotic event(s) (e.g., stroke, transient ischemic attacks, pulmonary embolism, deep vein thrombosis, or myocardial infarction) within 6 months of screening.
30. History or evidence of cardiac conditions, including congestive cardiac failure leading to marked limitation on physical activity, or inability to perform any physical activity without discomfort, ventricular arrhythmia requiring ongoing treatment, and atrial fibrillation.
31. Prior treatment with systemic anti-vascular endothelial growth factor (anti-VEGF) therapy.
32. Any concomitant or prior treatment with ethambutol (2 weeks prior to Day 1); deferoxamine and topiramate (4 weeks prior to Day 1); tamoxifen, hydroxychloroquine, chloroquine, or vigabatrin (8 weeks prior to Day 1), and amiodarone (12 weeks prior to Day 1).
33. Any investigational product administered for the treatment of neovascular Age-related Macular Degeneration prior to screening; and any investigational product (except dietary supplements, minerals or vitamins) for the treatment of ocular diseases or systemic diseases 30 days or 5 half-lives (whichever is longer), prior to screening, (see Table 5-1 for the list of prohibited medications).
34. Any prior or ongoing systemic medical condition (including but not limited to infectious, inflammatory, psychiatric, neurological, renal, hepatic, respiratory conditions or malignancies) or clinically significant screening laboratory value that in the opinion of the investigator may present a safety risk, interfere with study compliance and follow-up, or confound data interpretation throughout the study period.
35. Hypersensitivity to aflibercept, any of the excipients in SCB-420 or Eylea, or medications used during study procedures, (fluorescein, mydriatic eye drops, etc.), or any contraindication to study procedures or intravitreal injections, according to investigator judgment.
36. Any known allergy to povidone iodine or known serious allergy to the fluorescein sodium for injection in angiography.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular and non-ocular adverse events. | Baseline to Week 12
  Collection of any ocular and non-ocular adverse events.

SECONDARY OUTCOMES:
Change from baseline in Best Corrected Visual Acuity (BCVA) | Baseline to Week 12
  Change from baseline in Best Corrected Visual Acuity (BCVA)
Change in central foveal thickness (CFT) | Baseline to Week 12
  Change in central foveal thickness (CFT)
Percentage Change from baseline in the area of Choroidal neovascularization (CNV) lesions in Neovascular Age-related Macular Degeneration or polyps in Polypoidal choroidal vasculopathy | Baseline to Week 12
  Change in Choroidal neovascularization (CNV) lesions in Neovascular Age-related Macular Degeneration or polyps in Polypoidal choroidal vasculopathy
Observe serum concentration of free and total SCB 420 and Eylea | Baseline to Week 8
  Pharmacokinetic (PK) parameter area under the concentration versus time curves (AUC)
Observe maximum concentration (Cmax) of free and total SCB 420 and Eylea | Baseline to Week 8
  Pharmacokinetic (PK) parameter: Maximum concentration (Cmax)
Observe minimum concentration (Cmin) of free and total SCB 420 and Eylea | Baseline to Week 8
  Pharmacokinetic (PK) parameter: Minimum concentration (Cmin)
Observe Time to Maximum concentration (Tmax) of free and total SCB 420 and Eylea | Baseline to Week 8
  Description: Pharmacokinetic (PK) parameter: Time to maximum concentration (Tmax)
Observe Elimination Half Life (T1/2) of free and total SCB 420 and Eylea | Baseline to Week 8
  Pharmacokinetic (PK) parameter: Elimination Half Life (T1/2)
Titer of anti-drug antibodies (ADAs) against SCB-420 and Eylea at predose on Day 1, Week 4, and Week 8 | Baseline to Week 8
  Titer of anti-drug antibodies (ADAs) against SCB-420 and Eylea at predose on Day 1, Week 4, and Week 8
Neutralizing antibodies testing in confirmed ADA positive subjects | Baseline to Week 8
  Neutralizing antibodies testing in confirmed ADA positive subjects